CLINICAL TRIAL: NCT06932809
Title: Center Without Walls for Imaging Proteinopathies With PET (CW2IP2): Phase I Pilot Study of Biodistribution, Metabolism, Excretion and Brain Uptake of 18F-JSS20-183A
Brief Title: Study of Biodistribution, Metabolism, Excretion and Brain Uptake 18F-JSS20-183A
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 857138
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Tauopathies
Keywords: Positron Emission Tomography (PET); Brain MRI; Parkinsons Disease (PD); Alzheimers Disease (AD); Progressive Supranuclear Palsy (PSP); Corticobasal Syndrome (CBS); Genetic Frontotemporal Lobar Degeneration (Genetic FTLD)
MeSH Terms: conditions — Tauopathies; Parkinson Disease; Alzheimer Disease; Supranuclear Palsy, Progressive; Corticobasal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-JSS20-183A PET (Experimental): Participants will undergo 18F-JSS20-183A PET scan, they may also have a brain MRI and Amyloid PET scan as well as neurological assessments.
  Interventions: Drug: 18F-JSS20-183A PET; Diagnostic Test: Brain MRI; Diagnostic Test: Amyloid PET; Behavioral: Neurological Assessments

INTERVENTIONS:
Drug: 18F-JSS20-183A PET — 2 hour Positron Emission Tomography (PET) scan using new radiotracer 18F-JSS20-183A.
Diagnostic Test: Brain MRI — MRI scan of the brain.
Diagnostic Test: Amyloid PET — PET scan with Florbetaben F18 or 11C-PiB.
Behavioral: Neurological Assessments — Neurological assessments, including a video interview.

SUMMARY:
The current protocol is to determine the biodistribution, metabolism, excretion and brain uptake of 18F-JSS20-183A. The goal of this radiotracer is to quantify 4Repeat Tau (4Rtau) protein that is abnormally deposited in the brain of people with a class of neurodegenerative diseases called tauopathies, such as Progressive Supranuclear Palsy (PSP), Corticobasal Syndrome (CBS), syndromes of genetic Frontotemporal Lobar Degeneration (genetic FTLD) as well as participants with Parkinson disease (PD), Alzheimer's Disease (AD) and healthy controls. This multicenter project funded by an NIH U19 grant, is centered at U Pennsylvania (Penn, Grant PI: Robert Mach) in collaboration with U Pittsburgh (Pitt), Yale U, U of California at San Francisco (UCSF) and Washington University in St. Louis (WUSTL). The University of Pennsylvania will act as the sIRB for this multi-center human subjects project and participants will be recruited from all sites.

DETAILED DESCRIPTION:
The current protocol is to determine the biodistribution, metabolism, excretion and brain uptake of 18F-JSS20-183A. The goal of this radiotracer is to quantify 4Repeat Tau (4Rtau) protein that is abnormally deposited in the brain of people with a class of neurodegenerative diseases called tauopathies, such as Progressive Supranuclear Palsy (PSP), Corticobasal Syndrome (CBS), syndromes of genetic Frontotemporal Lobar Degeneration (genetic FTLD) as well as participants with Parkinson disease (PD), Alzheimer's Disease (AD) and healthy controls. This multicenter project funded by an NIH U19 grant, is centered at U Pennsylvania (Penn, Grant PI: Robert Mach) in collaboration with U Pittsburgh (Pitt), Yale U, U of California at San Francisco (UCSF) and Washington University in St. Louis (WUSTL). The University of Pennsylvania will act as the sIRB for this multi-center human subjects project and participants will be recruited from all sites.

Participating clinical sites will recruit up to 90 subjects total; up to 20 people with PSP, 10 with CBS, 15 with genetic FTLD, 10 with AD, 10 with PD and 25 healthy controls across sites with all participants ranging from 40-85 years old. We will encourage equal participation of males and females.

This protocol will include up to 90 evaluable participants across all centers (Penn, Yale, UCSF, WUSTL, Pitt), the whole-body biodistribution analysis will be done at Penn. Investigators anticipate enrollment of up to 15-20 participants at each clinical site, who will undergo up to 120-minutes of dynamic PET/CT scan over the brain, or brain and body if scanned on a long axial-field-of-view scanner, starting approximately at the same time as the injection of radiotracer. A second IV or an arterial line may be placed, preferably in the arm contralateral to the side of injection, for blood metabolite analysis and/or radioactive counts at various times during the scanning session. These blood sample collections can be omitted at the discretion of the investigator. For participants at Penn that may be part of BioD analysis, urine may be collected at the end of the scan session. Participants may also undergo a research brain MRI that may be on the same or a separate day from the PET.

PET imaging sessions will include an injection of ≤ 8 mCi (approximate range for most studies is anticipated to be 3-8 mCi at sites with a standard PET scanner or a lower dose may be used at sites with a high sensitivity scanner) of 18F-JSS20-183A. Biodistribution, metabolism, excretion and pilot brain uptake data will be collected and human dosimetry will be calculated from participants scanned at Penn who have whole body scans. PET scans will be collected to evaluate image quality and collect preliminary information on brain uptake of 18F-JSS20-183A in the disease cohorts and healthy controls. The safety of 18F-JSS20-183A will also be evaluated in all participants. Some participants (usually those with positive 18F-JSS20-183A PET scan) may also be asked to have an amyloid-beta (Aβ) PET scan or a blood draw to measure pTau to investigate specificity of 18F-JSS20-183A.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in all cohorts will be male or female adults from 40 to 85 years of age.
2. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures or Participants who are deemed unable to provide informed consent must have a designated study partner present for consent and to accompany them to study visits.

Investigators will ask disease cohort participants to agree to brain donation, but this choice is not mandatory for participation in this study.

Diagnosis-specific inclusion criteria: Clinical diagnoses will be determined by consensus committee (except AD and HC cohorts) for diagnostic agreement using video exams of each participant that are stored at WashU in a secured video repository with view-only access exclusively by secured virtual private network (VPN) connection. Video exam and screening assessments for PSP, CBS, MSA, PD, and FTLD may not be required to be repeated if they have been done within 6 months of enrollment, unless requested at the discretion of an investigator to document changes in clinical progression. A consensus committee will not be required to be repeated for participants who have already had a consensus committee diagnosis documented.

Exclusion Criteria:

1. Females who are pregnant or breast feeding will be excluded, a urine pregnancy test will be performed in women of child-bearing potential prior to injection of 18F-JSS20-183A 11C-PiB or 18F-Florbetaben
2. Forms of parkinsonism other than PSP-RS, and PD as defined above
3. History of significant or ongoing alcohol abuse or substance abuse or dependence based on medical record review or self-reported
4. Contraindications or inability to tolerate imaging, arterial line or IV placement or blood draw procedures in the opinion of an investigator or treating physician
5. Contraindication to MRI, such as non-compatible implanted medical device
6. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician or investigator to be a condition that could compromise participant safety or successful participation in the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Organ Biodistribution or Dosimetry | 4 weeks
  Determine biodistribution of the radioactive investigational drug, 18F-JSS20-183A and calculate human dosimetry. A second IV or an arterial line may be placed in the arm contralateral to the side of injection for blood metabolite analysis and/or radioactive counts at various times during the scanning session. Biodistribution, metabolism, excretion and pilot brain uptake data will be collected and human dosimetry will be calculated.
PET Uptake of Tracer | 4 weeks
  Determine whether there is selective uptake of 18F-JSS20-183A in people with taupathies compared to healthy volunteers and non-tau depositing neurodegenerative disease.

SECONDARY OUTCOMES:
Adverse Events | 4 weeks
  Adverse events will be collected.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California, San Francisco, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Early safety assessments including whole body dosimetry studies at Penn; coordinate patient selection criteria, centrally collect and serve all imaging and demographic data, coordinate tracer kinetic methods development and validation for human imaging, and coordinate all data to efficiently enable GO-NOGO decisions for candidate radiotracers. As a final check on diagnosis and specificity of candidate radiotracers, Investigators will request all patient participants to permit postmortem brain donation for autoradiography of relevant radiotracers on fresh frozen brain tissues. Additionally, this Core will interact with multiple ongoing studies with cohorts studying PD, MSA, PSP and FTD. Finally, a robust data sharing plan facilitates collaboration and use of support documents and imaging data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data shared as participants are enrolled and then final clinical report after study is completed.
Access Criteria: Dosimetry data. Dosimetry data for all compounds advanced to first-in-human trials will be provided on the website link for the Clinical Core. Since it is the intent of this U19 Center to provide information to the PET community on probes that have been validated in clinical research studies, these data will be provided once the CCOC has confirmed that a probe has met the validation criteria. This will include the results of dosimetry studies (organ, whole body, and EDE data) and, as requested, the organ radioactivity uptake, clearance curves and the dosimetry images in DICOM format.
  Imaging and Clinical Data. Links from the CCOC website will connect to XNAT and MARS to provide all de-identified clinical data, imaging data and related files including arterial blood sampling measurements. These data will be distributed upon request, as noted in the above policies for Data Sharing.